CLINICAL TRIAL: NCT04845308
Title: 3D Radiographic Evaluation of the Long Terms Results of Secondary Alveolar Bone Grafting in Patients With Alveolar Cleft: Comparison of Early Versus Late Secondary Grafting SABG : Secondary Alveolar Bone Grafting
Brief Title: Radiographic Evaluation of Secondary Alveolar Bone Grafting in Patients With Alveolar Cleft
Acronym: SABG
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0190
Record Dates: First submitted 2021-04-10; First posted 2021-04-14 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Alveolar Cleft
Keywords: Secondary alveolar bone grafting; 3D score; Navigation system; 3D-reconstruction; Bone loss
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Patients operated with an early secondary alveolar grafting between the ages of 4 to 7 years with a 3D imaging (CT, CBCT or scan) performed between the ages of 8 to 11 years.
- Group 2: Patients operated with a late secondary alveolar graft between the ages of 8 to 11 years with a 3D imaging (CT, CBCT or scan) performed at least 1 year after the operation.

SUMMARY:
Study about the comparison of post-operative results of secondary alveolar grafts according to two age groups: early secondary (4 to 7 years) versus late secondary (8 to 11 years) using a recently proposed score based on post-operative 3D CT analysis.

Comparison of the initial results of the graft in the two groups, with a reference 2D score and evaluation of the concordance between the results found with this score and those of the 3D score.

Finally, comparison of graft bone densities and nasal floor level (using 3D visualization) on post-operative TDMs in the 2 groups.

The aim of this study is to determine the optimal age for grafting using three-dimensional CT assessment.

ELIGIBILITY:
Inclusion criteria:

- Patients operated with an alveolar bone grafting for a single or bilateral labio-alveolar cleft in the pediatric plastic surgery department of the University Hospital of Montpellier between 1999 and 2021 and having had 3D imageries defined as:

* Group 1:

  o Patients operated with an early secondary alveolar grafting between the ages of 4 to 7 years with a 3D imaging (CT, CBCT or scan) performed between the ages of 8 to 11 years.
* Group 2:

  * Patients operated with a late secondary alveolar graft between the ages of 8 to 11 years with a 3D imaging (CT, CBCT or scan) performed at least 1 year after the operation.

Exclusion criteria:

* Patients operated with an alveolar bone grafting before 4 years or after 11 years
* Patients without post-operative CT

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients operated with an alveolar bone grafting (taken from the anterior iliac crest ) for a single or bilateral labio-alveolar cleft in the pediatric plastic surgery department of the University Hospital of Montpellier between 1999 and 2021.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Kamperos's score | Day 1
  Kamperos's score (a post-operative tri-dimensional scanographic score) This score includes 3 items measured on the post-operative CT: graft bone thickness (0 to 2), bone graft height (0 to 4) and nasal floor height (0 to 4).
  A total score of 0 to 8 is considered a failure and 9 to 10 a success

SECONDARY OUTCOMES:
Bergland's score | day 1
  Bergland's score (a post-operative two-dimensional radiographic score) Post-operative two-dimensional radiographic score : Use of the Bergland score (reference score).
  This score evaluates the height of the inter-dental bone septum up to the cemento - enamel junction (1 to 4).
Post-operative average bone density of the grafted area in axial slice | day 1
  Post-operative average bone density of the grafted area : in axial slice using radiological image processing software (Myrian®) to segment regions of interest.
Nasal floor level of the grafted side compared to the non grafted side using 3D visualization by volume rendering | day 1
  Nasal floor level by analyzing the level of the piriform orifice in relation to the grafted area using 3D visualization by volume rendering: percentage of the height between the piriform orifice to the alveolar crest of the grafted side relative to the controlateral side (the healthy side considered as the reference 100% side).

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume CAPTIER, MD.PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC